CLINICAL TRIAL: NCT05006950
Title: SPY Fluorescence Imaging Systems and Indocyanine Green to Determine the Percentage of Successful Critical Anatomy Recognition in Laparoscopic Cholecystectomy Surgeries.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business/strategic reasons and low accrual rate
Sponsor: Stryker Endoscopy (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CRD10283
Record Dates: First submitted 2021-08-09; First posted 2021-08-16 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Cholecystitis
MeSH Terms: conditions — Cholecystitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Stryker1688 Fluorescence imaging system — The purpose of this study is to use SPY fluorescence imaging systems and indocyanine green (ICG) as a tool to determine the percentage of successful critical anatomy recognition and to describe complications associated with intra-operative decision making in patients undergoing laparoscopic cholecystectomy.

SUMMARY:
This is a prospective single arm, single center study estimating percentage of successful critical anatomy recognition in laparoscopic cholecystectomy surgeries using SPY fluorescence imaging and ICG, with each surgery also providing a white light 360 degree images.

The primary objective is to determine the percentage of successful critical anatomy recognition using intra-operative SPY fluorescence imaging and ICG: and to describe complications associated with intra-operative decision making in patients undergoing laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age or older
* Subject is scheduled to undergo laparoscopic cholecystectomy, elective or emergent
* Subject provides informed consent and signs an approved informed consent document for the study
* Subject is willing to comply with the protocol and study visit schedule

Exclusion Criteria:

* Subject is pregnant or lactating
* Subject has a known allergy or history of adverse reaction to ICG, iodine or iodine dyes
* Subject has known history of cholangitis, pancreatitis, prior bile duct injury, coagulopathy or known pre-existing liver disease
* Subjects who, in the Investigator's opinion, have any medical condition that may make the subject a poor candidate for the investigation, interferes with the interpretation of study results, or integrity of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2022-02-08 (Actual); Study Completion 2022-09-07 (Actual)

PRIMARY OUTCOMES:
Outcome 1 | Intra-op visit
  To determine the percentage of successful critical anatomy recognition using intra-operative SPY fluorescence imaging and ICG in subjects undergoing laparoscopic cholecystectomy

SECONDARY OUTCOMES:
Outcome 2 | Intra-op visit
  To estimate the number of times a surgeon altered the surgical plan due to information identified/revealed by SPY fluorescence imaging

OTHER OUTCOMES:
Outcome 3 | Post op follow- up (7-14 days)
  To estimate the number of post-operative complications (related to gall bladder surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Anne Arundel Medical Center, Annapolis, Maryland, United States

IPD SHARING:
Plan to Share IPD: No